CLINICAL TRIAL: NCT03680443
Title: Total Hip Arthoplastry Revision by Dual-mobility Acetabular Cup Cemented in a Metal Reinforcement: A 62 Case Series at a Minimum 5 Years Follow-up
Brief Title: Total Hip Arthoplastry Revision by Dual-mobility Acetabular Cup Cemented in a Metal Reinforcement
Acronym: PTH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0041
Record Dates: First submitted 2018-08-21; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Aseptic Loosening; Arthroplasty Complications
Keywords: revision; reinforcement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assembly in THA revision — A single-center continuous series of 62 patients receiving such an assembly in THA revision was assessed retrospectively at a minimum 5 years' follow-up. Failure due to aseptic loosening or instability and implant survival at last follow-up were analyzed.

SUMMARY:
Total hip arthroplasty (THA) requires bone reconstruction in case of severe acetabular injury, with risk of dislocation, especially postoperatively. Dual-mobility cups have proved effective in preventing dislocation in THA revision for instability, but their behavior when cemented in a metal reinforcement has been little studied.

The present study assessed results for a dual-mobility cup cemented in a metal reinforcement, in terms of aseptic loosening and postoperative instability.

A single-center continuous series of 62 patients receiving such an assembly in THA revision was assessed retrospectively at a minimum 5 years' follow-up.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) requires bone reconstruction in case of severe acetabular injury, with risk of dislocation, especially postoperatively. Dual-mobility cups have proved effective in preventing dislocation in THA revision for instability, but their behavior when cemented in a metal reinforcement has been little studied.

The present study assessed results for a dual-mobility cup cemented in a metal reinforcement, in terms of aseptic loosening and postoperative instability.

A single-center continuous series of 62 patients receiving such an assembly in THA revision was assessed retrospectively at a minimum 5 years' follow-up. Failure due to aseptic loosening or instability and implant survival at last follow-up were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* patients between 19 and 84 years
* patients receiving such an assembly in THA revision

Exclusion Criteria:

* <19years
* > 94 years

Ages: 19 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 62 patients receiving such an assembly in THA revision was assessed retrospectively at a minimum 5 years' follow-up. Failure due to aseptic loosening or instability and implant survival at last follow-up were analyzed.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-04-26 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
dual-mobility cup cemented (effectiveness in terms of aseptic loosening) | 5 years
  The objective of the present study is to evaluate the most effective type of assembly , dual-mobility cup cemented in a metal reinforcement, in terms of aseptic loosening in the prevention of dislocation during the revision of the total hip arthroplasty (THA)

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Mertl, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No